CLINICAL TRIAL: NCT04400305
Title: "Increasing Physical Activity in Canadian Adults Who Have Been Affected by COVID-19 Social Distancing Restrictions: A Feasibility Trial of an Online Intervention"
Brief Title: "Increasing Physical Activity in Canadian Adults Affected by COVID-19 Social Distancing Restrictions: A Feasibility Trial of an Online Intervention"
Acronym: COVID-19
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Victoria (Other)
Responsible Party: Principal Investigator, Ryan Rhodes, Professor Ryan Rhodes, University of Victoria
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 05-281983
Record Dates: First submitted 2020-05-21; First posted 2020-05-22 (Actual); Last update posted 2021-10-21 (Actual); Status verified 2021-10

CONDITIONS: Physical Activity, Healthy Promotion
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): No Intervention: Control Group This group will complete baseline and final questionnaires (online). At the end of the study this group will have the option to receive access to the other group's materials (online platform) if they wish, for the 6 week period following the study.
- Intervention (Other): Participants will complete a baseline questionnaire, and receive access to the our online platform for 6 weeks. Completing the online platform is designed to encourage participants to engage in physical activity. At 3 weeks, a check-in session will occur over the phone. At 6 weeks the participant will be contacted to complete the final questionnaire, and do a wrap up interview. The end-of-trial qualitative interview will evaluate participant satisfaction and feasibility of the intervention. For this reason a lab employee unaffiliated with this study will complete these in person interviews.
  Interventions: Behavioral: Digital Health Online Platform

INTERVENTIONS:
Behavioral: Digital Health Online Platform — The website has 10 lessons that the participant will gain access to on a bi-weekly basis. Lesson titles are as follows:
  Lesson 1 - Benefits of Physical Activity on Chronic Disease Lesson 2 - Mental benefits of Physical Activities Lesson 3 - Increasing Self Confidence for Physical Activities Lesson 4 - Learning about your Emotions Lesson 5 - Building Social Support Lesson 6 - Building Physical Activity Opportunity Lesson 7 - Goal Setting and Planning Lesson 8 - Self Monitoring Lesson 9 - Habit Lesson 10 - Identity
  Arms: Intervention

SUMMARY:
Internet-based health promotion programs have the potential to reach more individuals than in person interventions, without overtaxing healthcare resources. Having a high quality, user-centered web-based program can help maximize user engagement and adherence. Thus, the primary objective of this pilot study is to examine the feasibility, time, cost, and acceptability of a web-based physical activity behavior change program with Canadian Adults who have had to start practising/following the social distancing guidelines due to the COVID-19 situation. We will also be examining changes other behavioral indicators related to PA as a secondary outcome measure.

DETAILED DESCRIPTION:
Background: Physical activity is associated with management and/or prevention of over 25 chronic health conditions; however the majority of adults in North America are not active enough to experience these benefits. Behavioral strategies have been shown to be effective for increasing physical activity, and our online platform includes components of several behavioral strategies including goal setting and feedback.

Target Population: Participants will be Canadian adults over 18 who have

1. recently started practising social distancing due to our current COVID-19 situation
2. currently are participating in physical activity below Canadian recommended guidelines (150 minutes of moderate to vigorous activity per week).
3. Participants must have access to the Internet. Sample Size: 40 participants, 20 participants per group - (Control) 20 participants (intervention) Participants will be excluded from the project if they do not have access to the Internet, are unable to speak/read English, are not engaging in moderate-to vigorous PA (MVPA) sufficient to meet the PA Guidelines, have an existing chronic medical condition potentially making them at risk of injury or ill health from increasing their physical activity (assessed using the GAQ. Screening will be completed formally over the phone, and participants will give their consent online.

Condition one: Waitlist control group: One group (evenly representing Adults practising social distancing) will complete the baseline and final questionnaires (online). At the end of the study this group will have the option to receive access to the other group's materials (online platform) if they wish, for the 6 week period following the study. Access to the online platform is for study participant use and benefit only and no participant data/website analytics will be collected at this point in the study.

Condition two: One group (evenly representing Adults practising social distancing) will complete the online baseline questionnaire, and receive access to the online platform. Briefly, the participants will be shown (via skype, Face time, Zoom or other alternate online technology) how to use it .

At 3 weeks, a check-in session will occur, depending on what the participant prefers, a researcher will arrange a virtual visit or phone call with the participant to chat about how their physical activity has been going and to ensure the web application' usability. Again at this point on-going consent will be secured. At 6 weeks a researcher will arrange a virtual visit or phone call with the participant & ask them to complete the final online questionnaire and do a wrap up interview. The end-of-trial qualitative interview will evaluate participant satisfaction and feasibility of the intervention. For this reason a lab employee unaffiliated with this study will complete these interviews via skype or alternate technology. The interview will be audio-recorded transcribed verbatim. After the intervention group participants have completed the 6 week online program, data collection will be complete and while they may still access the platform for an additional 6 weeks, data collection from participants or website use analytics will not be ongoing.

ELIGIBILITY:
Inclusion Criteria:

Potential participants will be included if they have:

1. started practising social distancing due to the current COVID-19 guidelines
2. are currently not meeting the physical activity (PA) guidelines (less than 150 minutes of moderate to vigorous aerobic activity)
3. participants must have access to the internet at home, and have a smart phone or home computer that can support the eHealth application we are using.

Exclusion Criteria:

Participants will be excluded from the project if:

1. they do not have access to the Internet,
2. are unable to speak/read English,
3. are engaging in moderate-to vigorous PA (MVPA) sufficient to meet the PA Guidelines,
4. have an existing chronic medical condition potentially making them at risk of injury or ill health from increasing their physical activity (this will be assessed using the GAQ. Screening completed formally over the phone, and participants will give their consent online)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2020-05-20 (Actual); Primary Completion 2021-08-30 (Actual); Study Completion 2021-08-30 (Actual)

PRIMARY OUTCOMES:
Recruitment rate (monthly) | 4 months
  For the full scale RCT, we are looking for a 1 day per week or 30 min MVPA change which equates to an approximate effect size of d = .35. This equates to roughly 65 per group (130 for a two group trial). If we recruit for 2 years in the large trial (assuming a six month time period for each person in the intervention) we need to be recruiting at least 6 per month.
Participant retention | 6 weeks
  Number of participants who complete both baseline and end of study (6 week) measures. A 80-100% retention rate is indicative of a strong trial (Jackson & Waters, 2005).
Participant intervention satisfaction/evaluation | 6 Weeks
  For satisfaction ratings, mean and standard deviations will be calculated for the quantitative satisfaction and evaluation questionnaire. Given that scores of 1 (ex. not helpful, did not use the tools) and 2 (ex. Somewhat helpful, used a little bit of the tools) indicated levels of dissatisfaction, and 3 (ex. Quite helpful, used a bit of the tools) and 4 (ex. Extremely helpful, used a lot of the tools) indicated some sort of satisfaction, a mean score of ≥ 2.5 will be deemed acceptable for recommendation for a full RCT.

SECONDARY OUTCOMES:
Change in self-reported physical activity from baseline to 6 weeks | 6 Weeks
  Measured from questionnaire using Godin's personal self report leisure time measurement tool, also known as the Leisure Score Index (LSI). The Leisure Score Index contains three questions, which assess the frequency of mild, moderate, and strenuous activity performed for at least 10 minutes during free time in a typical week. Changes in these measures will be examined
Change in physical activity beliefs, attitudes, barriers, and motivation from baseline to 6 weeks. | Baseline - 6 weeks
  Included in questionnaire - Ajzen's theory of planned behaviour questionnaire will be applied to measure participants' beliefs, attitudes, barriers, and motivation related to physical activity.
Change in physical activity behaviour regulation from baseline to 6 weeks. | Baseline - 6 weeks
  Included in questionnaire - 5 items adapted from Umstattd's scale measuring physical activity self-regulation strategies. Changes in this measure will be examined. The Behavioural Regulation in Exercise Questionnaire - 5 point Likert Scale 1 = Strongly agree to 5 = Strongly Disagree
Change in physical activity habits from baseline to 6 weeks | Baseline - 6 weeks
  Included in questionnaire - 12 Self Report Habit Index items from the measure developed by Verplanken and Orbell and adapted to physical activity by Chatzisarantis and Hagger. Changes in this measure will be examined. Physical Activity Participation Habits Questionnaire - Habit Index - 5 point Likert Scale 1 = Strongly agree to 5 = Strongly Disagree
Change in physical activity identity from baseline to 6 weeks | Baseline - 6 weeks
  Included in questionnaire - Anderson and Cychosz Exercise Identity Scale is used to measure participants' identification as someone who participates in physical activity. Physical Activity Participation Identity Questionnaire - Identity Scale - 5 point Likert Scale 1 = Strongly agree to 5 = Strongly Disagree
Change in life satisfaction measured using the Short Form 12 questionnaire from baseline to 6 weeks | Baseline - 6 weeks
  Change in life satisfaction from baseline to 6 weeks measured using Diener's satisfaction with life scale in a questionnaire.
  The online questionnaire will asses participants' life satisfaction using Diener's satisfaction with life scale. Changes in this measure will be examined (6 weeks to baseline) [Time Frame: Baseline to 6 weeks] Variable scale.

CONTACTS AND LOCATIONS:
Locations (2):
- Canada (2):
  - Behavioural Medicine Lab, University of Victoria, Victoria, British Columbia
  - University of Victoria, Victoria, British Columbia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jackson N, Waters E; Guidelines for Systematic Reviews in Health Promotion and Public Health Taskforce. Criteria for the systematic review of health promotion and public health interventions. Health Promot Int. 2005 Dec;20(4):367-74. doi: 10.1093/heapro/dai022. Epub 2005 Sep 16. PMID 16169885